CLINICAL TRIAL: NCT00787332
Title: A Comparative Clinical and Pharmacoeconomic Study Comparing Argatroban® IV vs Desirudin SC for Patients With Suspected Heparin-Induced Thrombocytopenia (HIT)With or Without Thrombosis Syndrome (HIT/TS)
Brief Title: A Comparative Sudy Comparing Argatroban® IV vs Desirudin SC for Suspected HIT With or Without Thrombosis Syndrome
Acronym: HIT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Canyon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DES-08-01
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Results first posted 2012-12-31 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Suspected Heparin-Induced Thrombocytopenia
Keywords: Suspected Heparin Induced Thrombocytopenia (HIT)
MeSH Terms: interventions — desirudin; argatroban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desirudin (Experimental): Patients with suspected HIT without thrombosis syndrome (HIT/TS), randomized to SC Desirudin
  Interventions: Drug: Desirudin or Argatroban®
- Argatroban® (Active Comparator): Patients randomized to IV Argatroban®
  Interventions: Drug: Desirudin or Argatroban®

INTERVENTIONS:
Drug: Desirudin or Argatroban® — Desirudin 15mg SC Argatroban® IV dosing per Package Insert

SUMMARY:
Compare Clinical Success and Costs in two Arms

DETAILED DESCRIPTION:
Demonstrate clinical and economic utility between the study Arms.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written Informed Consent
2. Be at least 18 years of age.
3. A suspicion of heparin-induced thrombocytopenia with or without thrombosis syndrome (HIT/TS) due to one of the following clinical scenarios:

   1. Patients who are receiving heparin/LMWH or have received heparin/LMWH within the previous 100 days AND one of the following:

      * have a fall in platelet count of > 30% from a baseline prior to heparin/LMWH, OR
      * have a thrombotic event, OR
      * develop skin lesions secondary to subcutaneous heparin (even if the patient is no longer receiving heparin therapy when thrombocytopenia, thrombosis or skin lesions occur).

      Patients with thrombosis or skin lesions need not have concomitant thrombocytopenia to be included.
   2. A rapid fall in the platelet count by >30% from baseline within 24 hours after starting heparin/LMWH in patients with suspected exposure to heparin or LMWH in the previous 100 days (e.g. hospitalization or invasive procedure within the past 100 days).
   3. In post-operative cardiac surgery patients, development of thrombocytopenia defined as a decrease in platelet count by >30% from the post-operative peak; or patients whose platelet count fails to increase post-operatively (e.g. remains < 100,000 mm3 at Day 4 or later, calendar day of surgery=Day 0).
4. In patients with the diagnosis of HIT/TS established by a hematology consultant, but in whom the above criteria are not fulfilled, the Investigator should contact the Medical Monitor for consideration of the patient's inclusion in this study (A hematology consult is highly advisable, but not required prior to randomization).

Exclusion Criteria:

* Confirmed pregnancy (if woman of child-bearing potential- urine or serum pregnancy test).
* Patients with suspected or confirmed pulmonary embolism, requiring continued anticoagulation or acute ischemic stroke will be excluded
* Cerebrovascular accident within the previous 6 months
* Intracranial neoplasm, arteriovenous malformation or aneurysm.
* Severe renal insufficiency as determined by measured or estimated creatinine clearance < 30 ml/min.
* Known allergy to Argatroban®, Desirudin or hirudin derived drugs, or known sensitivity to any component of the product
* Patients receiving recombinant hirudin (e.g. lepirudin) within the previous 6 months prior to enrollment.
* Patients receiving >2 doses of fondaparinux for treatment of suspected HIT
* Multi-system organ failure or estimated survival of less than 30 days.
* Participation in other clinical research studies involving the evaluation of other investigational drugs or devices within 30 days of enrollment
* Refusal to undergo blood transfusion should it become necessary
* Active bleeding or irreversible coagulation abnormality
* Uncontrolled hypertension defined as a blood pressure >180/110 mm Hg.
* Patients requiring indwelling mechanical intervention such as left-ventricular assist device, intra-aortic balloon pump, veno-venous ultra filtration, etc.
* Severe liver disease and any other disease or condition, which, in the judgment of the Investigator, would place a patient at undue risk by being enrolled in the trial, or cause inability to comply with the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Bell, PharmD, Study Director — Canyon Pharmaceuticals, Inc.
Locations (24):
- United States (24):
  - University of Colorado Health Science Center, Aurora, Colorado
  - Washington Regional Cardiac Surgery, Washington D.C., District of Columbia
  - Florida Hospital Cardiovascular Research, Orlando, Florida
  - University of South Florida, Tampa General Hospital, Tampa, Florida
  - Emory University, Emory Crawford Long Hospital, Atlanta, Georgia
  - Kaiser Permanente Medical Center, Honolulu, Hawaii
  - Provena St. Joseph's Medical Center, Joliet, Illinois
  - Mercy Medical Center, Sioux City, Iowa
  - Maine Medical Center, Portland, Maine
  - William Beaumont Hospital, Royal Oak, Michigan
  - St Mary's Hospital Rochester, Mayo Clinic, Rochester, Minnesota
  - UMDNJ-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - St Vincent's Hosptial -Manhattan, Manhattan, New York
  - Mount Sinai Clinical & Translational Research Institute, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, Moses Division, The Bronx, New York
  - Forsyth Regional Medical Center, Winston-Salem, North Carolina
  - The Cleveland Clinic, Cleveland, Ohio
  - Cardiothoracic Vascular Surgial Specialists, Columbus, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Methodist Hospital, Houston, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Charleston Area Medical Center, Charleston, West Virginia

REFERENCES:
- [Derived] Boyce SW, Bandyk DF, Bartholomew JR, Frame JN, Rice L. A randomized, open-label pilot study comparing desirudin and argatroban in patients with suspected heparin-induced thrombocytopenia with or without thrombosis: PREVENT-HIT Study. Am J Ther. 2011 Jan;18(1):14-22. doi: 10.1097/MJT.0b013e3181f65503. PMID 21079512
- [Derived] Frame JN, Rice L, Bartholomew JR, Whelton A. Rationale and design of the PREVENT-HIT study: a randomized, open-label pilot study to compare desirudin and argatroban in patients with suspected heparin-induced thrombocytopenia with or without thrombosis. Clin Ther. 2010 Apr;32(4):626-36. doi: 10.1016/j.clinthera.2010.04.012. PMID 20435232

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between November 2008 and December 2009 from approximately 20 US Medical Centers
Pre-assignment Details: Patients were excluded if they had severe renal failure (CrCL<30 mL/min), known allergy to r-hirudins or argatroban, multisystem organ failure, uncontrolled bleeding.
Groups:
- Desirudin: Patients with suspected HIT randomized to SC Desirudin in a 1:1 ratio
- Argatroban®: Patients with suspected HIT randomized to IV Argatroban® in a 1:1 ratio
Period: Overall Study
Arm/Group | Desirudin | Argatroban®
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Desirudin: Patients with suspected HIT randomized to SC Desirudin i
- Argatroban®: Patients with suspected HIT randomized to IV Argatroban®
- Total: Total of all reporting groups
Arm/Group | Desirudin | Argatroban® | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 2 | 2 | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 69 (9.5) | 62 (9.3) | 65 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: New Thrombosis, Amputation, Death, Major and Minor Bleeding
Time Frame: 30 days
Population: All patients receiving drug
Measure: Number; unit: participants
Arm/Group | Desirudin | Argatroban®
Number analyzed (Participants) | 8 | 8
participants | 1 | 5

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Desirudin | Argatroban®
Serious Adverse Events (participants affected / at risk) | 1/8 | 2/8
Other Adverse Events (participants affected / at risk) | 7/8 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desirudin (N=8) | Argatroban® (N=8)
esophageal hematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sublingual Hematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
femoral graft thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desirudin (N=8) | Argatroban® (N=8)
leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
non-sustained ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
right groin hematoma (Vascular disorders) | 0 (0) | 1 (1)
anxiety (Nervous system disorders) | 1 (1) | 0 (0)
sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
elevated LFT's (Gastrointestinal disorders) | 2 (2) | 1 (1)
mild rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
shingles (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
fever (Infections and infestations) | 1 (1) | 0 (0)
clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study stopped early due to poor enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No